CLINICAL TRIAL: NCT04620369
Title: Rose Geranium in Sesame Oil Nasal Spray as an Agent to Improve Symptoms of Nasal Vestibulitis: A Phase III Double Blinded Randomized Controlled Trial
Brief Title: Rose Geranium in Sesame Oil Nasal Spray for the Improvement of Nasal Vestibulitis Symptoms in Cancer Patients Receiving Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MC19C1; NCI-2020-08287 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-10-27; First posted 2020-11-09 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2023-10

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Nasal Vestibulitis
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (rose geranium in sesame oil nasal spray) (Experimental): Patients instill rose geranium in sesame oil nasal spray, 1 spray in each nostril BID on days 1-14 in the absence of unacceptable toxicity.
  Interventions: Other: Questionnaire Administration; Drug: Rose Geranium in Sesame Oil Nasal Spray
- Arm B (isotonic nasal saline) (Placebo Comparator): Patients instill isotonic nasal saline, 1 spray in each nostril BID on days 1-14 in the absence of unacceptable toxicity. After 2 weeks, patients may instill rose geranium in sesame oil nasal spray as in Arm A for an additional 2 weeks in the absence of unacceptable toxicity.
  Interventions: Drug: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Placebo Administration — Instill isotonic nasal saline intranasally
  Arms: Arm B (isotonic nasal saline)
Other: Questionnaire Administration — Ancillary studies
Drug: Rose Geranium in Sesame Oil Nasal Spray — Instill intranasally
  Arms: Arm A (rose geranium in sesame oil nasal spray)

SUMMARY:
This phase III trial compares rose geranium in sesame oil nasal spray to isotonic nasal saline in improving symptoms of nasal vestibulitis in cancer patients receiving chemotherapy. Nasal (nose) symptoms (dryness, discomfort, bleeding, scabbing or sores) due to inflammation, termed nasal vestibulitis, is reported as a side effect of cancer-directed therapy. Rose geranium in sesame oil nasal spray may work better than isotonic nasal saline in improving symptoms of nasal vestibulitis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the ability of rose geranium in sesame oil nasal spray to alleviate nasal vestibulitis in patients undergoing systemic, antineoplastic therapy when compared with isotonic nasal saline.

SECONDARY OBJECTIVE:

I. To assess toxicities related to rose geranium in sesame oil nasal spray in this study situation.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients instill rose geranium in sesame oil nasal spray, 1 spray in each nostril twice daily (BID) on days 1-14 in the absence of unacceptable toxicity.

ARM B: Patients instill isotonic nasal saline, 1 spray in each nostril BID on days 1-14 in the absence of unacceptable toxicity. After 2 weeks, patients may instill rose geranium in sesame oil nasal spray as in Arm A for an additional 2 weeks in the absence of unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* REGISTRATION-INCLUSION CRITERIA
* Age >= 18 years and be diagnosed with cancer and receiving chemotherapy
* Ability to provide informed consent
* Willingness to complete questionnaires
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, 2
* One or more of the following nasal symptoms for which the patient reports they would appreciate treatment. Symptoms must have started after the initiation of systemic, antineoplastic therapies, be attributed to the systemic, antineoplastic therapies, and symptoms must be reported as being moderate (corresponding to a score of 2) or worse on a scale from mild (1) to very severe (4) on at least one of the items below.

  * Dryness
  * Discomfort/pain
  * Bleeding
  * Scabbing
  * Sores

Exclusion Criteria:

* REGISTRATION-EXCLUSION CRITERIA
* Predisposition to epistaxis prior to the initiation of cancer-directed therapy (more than once a month over the previous year)
* Planned initiation or continuation of any topical nasal treatment other than the studied nasal spray,(such as nasal steroids, Ayr nasal gel, Neosporin ointment or nasal administration of petroleum jelly). Taking Imitrex for migraines is acceptable
* Previous exposure to rose geranium in sesame oil nasal spray
* Concurrent upper respiratory tract infection
* History of allergic or other adverse reactions to sesame oil or essential rose geranium oil
* Any other reason that the study clinician or investigator feels precludes safe or appropriate inclusion in this study
* Vulnerable populations: pregnant women, prisoners, mentally handicapped
* RE-REGISTRATION
* The patient will be un-blinded and determined to have been on the saline arm, when initially randomized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles L Loprinzi, Principal Investigator — Mayo Clinic in Rochester
Locations (20):
- United States (20):
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Ely Clinic, Ely, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Fairview Grand Itasca Clinic & Hospital, Grand Rapids, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Range Medical Center, Hibbing, Minnesota
  - Essentia Health - International Falls Clinic, International Falls, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota

REFERENCES:
- [Derived] Cathcart-Rake EJ, Steinert K, Smith D, Lewis-Peters S, Giridhar K, Novotny P, Dauer D, O'Connor A, Thome S, Erickson MK, Friday BB, Loprinzi CL. Rose geranium in sesame oil nasal spray to improve nasal vestibulitis symptoms: a randomized controlled trial. Support Care Cancer. 2024 May 24;32(6):379. doi: 10.1007/s00520-024-08580-6. PMID 38789656

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 patients on Arm A did crossover despite the protocol saying otherwise
Groups:
- Arm A (Rose Geranium in Sesame Oil Nasal Spray): Patients instill rose geranium in sesame oil nasal spray, 1 spray in each nostril BID on days 1-14 in the absence of unacceptable toxicity.
  >>
  >
  >>
  >>
  >
  >> Questionnaire Administration: Ancillary studies
  >>
  >
  >>
  >>
  >
  >> Rose Geranium in Sesame Oil Nasal Spray: Instill intranasally
- Arm B (Isotonic Nasal Saline): Patients instill isotonic nasal saline, 1 spray in each nostril BID on days 1-14 in the absence of unacceptable toxicity. After 2 weeks, patients may instill rose geranium in sesame oil nasal spray as in Arm A for an additional 2 weeks in the absence of unacceptable toxicity.
  >>
  >
  >>
  >>
  >
  >> Placebo Administration: Instill isotonic nasal saline intranasally
  >>
  >
  >>
  >>
  >
  >> Questionnaire Administration: Ancillary studies
Period: Initial Study
Arm/Group | Arm A (Rose Geranium in Sesame Oil Nasal Spray) | Arm B (Isotonic Nasal Saline)
Started | 53 | 53
Completed | 52 | 50
Not Completed | 1 | 3
Period: Crossover
Arm/Group | Arm A (Rose Geranium in Sesame Oil Nasal Spray) | Arm B (Isotonic Nasal Saline)
Started | 2 | 37
Completed | 2 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A (Rose Geranium in Sesame Oil Nasal Spray); Arm B (Isotonic Nasal Saline): Patients instill rose geranium in sesame oil nasal spray, 1 spray in each nostril BID on days 1-14 in the absence of unacceptable toxicity.> >>>
  >
  >>> Questionnaire Administration: Ancillary studies>
  >>>
  >
  >>> Rose Geranium in Sesame Oil Nasal Spray: Instill intranasally
- Total: Total of all reporting groups
Arm/Group | Arm A (Rose Geranium in Sesame Oil Nasal Spray) | Arm B (Isotonic Nasal Saline) | Total
Number analyzed (Participants) | 43 | 41 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (12.3) | 59.3 (12.3) | 59.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 37 | 73
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 43 | 40 | 83
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 40 | 40 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Prior treatments for nose symptoms [Count of Participants; unit: Participants]
  0 | 32 | 25 | 57
  1 | 7 | 11 | 18
  2 | 2 | 5 | 7
  3+ | 2 | 0 | 2
Prior history of allergies or asthma [Count of Participants; unit: Participants] | 16 | 15 | 31
Currently smoking [Count of Participants; unit: Participants]
  No | 36 | 37 | 73
  Yes | 7 | 4 | 11
Taking aspirin or blood thinners [Count of Participants; unit: Participants] | 8 | 6 | 14
Most bothersome nasal symptom [Count of Participants; unit: Participants]
  Dryness | 15 | 15 | 30
  Discomfort | 7 | 4 | 11
  Bleeding | 19 | 10 | 29
  Scabbing | 0 | 7 | 7
  Sores | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Response
Description: Response is determined from a patient global impression of change scale and is defined as a patient reporting that the nasal symptom that was most prominent prior to starting the study has been moderately better or very much better 2 weeks after initiating the nasal spray. The number and percentage of patients experiencing a response 2 weeks after initiating>>> the nasal spray will be estimated within each randomized arm and the corresponding two-sided 95% exact (Clopper-Pearson) confidence interval provided. A between-arm comparison of the proportion of patients experiencing a response 2 weeks after initiating the nasal spray will be made using the Fisher's exact test.
Time Frame: At 2 weeks after initiating the nasal spray
Measure: Count of Participants; unit: Participants
Groups:
- Arm A (Rose Geranium in Sesame Oil Nasal Spray): Patients instill rose geranium in sesame oil nasal spray, 1 spray in each nostril BID on days 1-14 in the absence of unacceptable toxicity.>>> >>> Questionnaire Administration: Ancillary studies>>>
  >>> Rose Geranium in Sesame Oil Nasal Spray: Instill intranasally
- Arm B (Isotonic Nasal Saline): Patients instill isotonic nasal saline, 1 spray in each nostril BID on days 1-14 in the absence of unacceptable toxicity. After 2 weeks, patients may instill rose geranium in sesame oil nasal spray as in Arm A for an additional 2 weeks in the absence of unacceptable toxicity.>>> >>> Placebo Administration: Instill isotonic nasal saline intranasally>>>
  >>> Questionnaire Administration: Ancillary studies
Arm/Group | Arm A (Rose Geranium in Sesame Oil Nasal Spray) | Arm B (Isotonic Nasal Saline)
Number analyzed (Participants) | 43 | 41
Participants
  worsening of nasal symptoms | 2 | 4
  no change | 1 | 12
  some nasal symptom improvement | 40 | 25

2. Secondary Outcome: Severity of Most Prominent Nasal Symptom Indicated at Baseline
Description: For the most prominent nasal symptom indicated at baseline, patients will record the severity on an ordinal scale of 1=mild, 2=moderate, 3=severe, and 4=very severe. Two weeks after initiating the nasal spray the patients will record the severity of the most prominent nasal symptom as 0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe. A shift table will be created to descriptively display the number of patients who record a 1, 2, 3, or 4 at baseline and the shift two-weeks after initiating the nasal spray. In addition, the within-patient change in severity of the most prominent nasal symptom will be calculated 2 weeks after initiating the nasal spray and summarized descriptively within each arm. The Wilcoxon rank-sum test will be performed, and the methods of Hodges and Lehmann will be applied to compute a point estimate and confidence interval for the difference in medians between the two arms.
Time Frame: Up to 2 weeks after initiating the nasal spray
Measure: Mean (Standard Deviation); unit: "percentage of Week 0 score
Groups:
- Arm A (Rose Geranium in Sesame Oil Nasal Spray): Patients instill rose geranium in sesame oil nasal spray, 1 spray in each nostril BID on days 1-14 in the absence of unacceptable toxicity.
  >>>
  >>> Questionnaire Administration: Ancillary studies
  >>>
  >>> Rose Geranium in Sesame Oil Nasal Spray: Instill intranasally
- Arm B (Isotonic Nasal Saline): Patients instill isotonic nasal saline, 1 spray in each nostril BID on days 1-14 in the absence of unacceptable toxicity. After 2 weeks, patients may instill rose geranium in sesame oil nasal spray as in Arm A for an additional 2 weeks in the absence of unacceptable toxicity.
  >>>
  >>> Placebo Administration: Instill isotonic nasal saline intranasally
  >>>
  >>> Questionnaire Administration: Ancillary studies
Arm/Group | Arm A (Rose Geranium in Sesame Oil Nasal Spray) | Arm B (Isotonic Nasal Saline)
Number analyzed (Participants) | 43 | 41
"percentage of Week 0 score
  Week 0 | 100 (0) | 100 (0)
  Week 1 | 70.155 (4.520) | 91.458 (5.598)
  Week 2 | 65.0 (5.154) | 77.724 (4.890)

3. Secondary Outcome: Nasal Symptom Analysis
Description: Each nasal symptom (dryness, pain, bleeding, and scabbing) will be descriptively summarized, tabulated, and plotted according to arm at baseline, and at 1 and 2 weeks post-baseline; additionally, will group patients according to baseline severity for each symptom and summarize changes over time and according to arm. Shift tables will also be generated to descriptively display the number of patients who record a 1, 2, 3, or 4 at baseline and the shift one- and two-weeks after initiating the nasal spray. The Nasal symptom scale is 0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe with very severe being the worst outcome.
Time Frame: Up to 2 weeks after initiating the nasal spray
Population: Some patients missed their post-baseline assessment
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Arm A (Rose Geranium in Sesame Oil Nasal Spray): Patients instill rose geranium in sesame oil nasal spray, 1 spray in each nostril BID on days 1-14 in the absence of unacceptable toxicity.
  >>
  >> Questionnaire Administration: Ancillary studies
  >>
  >> Rose Geranium in Sesame Oil Nasal Spray: Instill intranasally
- Arm B (Isotonic Nasal Saline): Patients instill isotonic nasal saline, 1 spray in each nostril BID on days 1-14 in the absence of unacceptable toxicity. After 2 weeks, patients may instill rose geranium in sesame oil nasal spray as in Arm A for an additional 2 weeks in the absence of unacceptable toxicity.
  >>
  >> Placebo Administration: Instill isotonic nasal saline intranasally
  >>
  >> Questionnaire Administration: Ancillary studies
Arm/Group | Arm A (Rose Geranium in Sesame Oil Nasal Spray) | Arm B (Isotonic Nasal Saline)
Number analyzed (Participants) | 43 | 41
score on a scale
  Dryness Week 0 | 2.95 [2.68 to 3.23] | 3.14 [2.91 to 3.39]
  Dryness Week 1: number analyzed (Participants) | 43 | 40
  Dryness Week 1 | 2.02 [1.79 to 2.26] | 2.8 [2.56 to 3.04]
  Dryness Week 2 | 2 [1.72 to 2.28] | 2.46 [2.15 to 2.77]
  Tenderness/Discomfort Week 0 | 2.63 [2.29 to 2.96] | 2.46 [2.14 to 2.79]
  Tenderness/Discomfort Week 1: number analyzed (Participants) | 43 | 40
  Tenderness/Discomfort Week 1 | 1.65 [1.40 to 1.90] | 2.25 [1.91 to 2.59]
  Tenderness/Discomfort Week 2: number analyzed (Participants) | 42 | 41
  Tenderness/Discomfort Week 2 | 1.67 [1.38 to 1.96] | 1.98 [1.64 to 2.31]
  Bleeding Week 0 | 2.56 [2.24 to 2.88] | 2.68 [2.36 to 3.00]
  Bleeding Week 1: number analyzed (Participants) | 43 | 40
  Bleeding Week 1 | 2 [1.69 to 2.31] | 2.48 [2.18 to 2.77]
  Bleeding Week 2 | 1.72 [1.42 to 2.02] | 2 [1.71 to 2.29]
  Scabbing Week 0 | 2.72 [2.40 to 3.05] | 2.49 [2.13 to 2.84]
  Scabbing Week 1: number analyzed (Participants) | 43 | 40
  Scabbing Week 1 | 1.74 [1.48 to 2.00] | 2.25 [1.95 to 2.55]
  Scabbing Week 2 | 1.63 [1.36 to 1.90] | 2.17 [1.83 to 2.52]
  Sores Week 0 | 2.14 [1.84 to 2.44] | 1.93 [1.59 to 2.27]
  Sores Week 1: number analyzed (Participants) | 43 | 40
  Sores Week 1 | 1.58 [1.32 to 1.84] | 1.8 [1.51 to 2.09]
  Sores Week 2 | 1.47 [1.21 to 1.72] | 1.78 [1.48 to 2.08]
  Most Prominent Symptom Week 0 | 3.09 [2.82 to 3.37] | 3.17 [2.92 to 3.42]
  Most Prominent Symptom Week 1: number analyzed (Participants) | 43 | 40
  Most Prominent Symptom Week 1 | 2.09 [1.79 to 2.39] | 2.73 [2.46 to 2.99]
  Most Prominent Symptom Week 2: number analyzed (Participants) | 42 | 41
  Most Prominent Symptom Week 2 | 1.93 [1.63 to 2.22] | 2.39 [2.09 to 2.69]

4. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The constellation of AEs as scored using the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 will be summarized within arms by reporting the number and percentage of patients. Specifically, to evaluate the AE profiles associated with each arm, the maximum grade for each type of AE will be recorded for each patient and frequency tables will be reviewed to determine overall patterns and compared between arms using Wilcoxon tests.
Time Frame: Up to 2 weeks after initiating the nasal spray
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Rose Geranium in Sesame Oil Nasal Spray) | Arm B (Isotonic Nasal Saline)
Number analyzed (Participants) | 43 | 41
Participants
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 weeks
Groups:
- Arm B (Isotonic Nasal Saline); Arm A Crossover; Arm B Crossover: Rose Geranium in Sesame Oil Nasal Spray: Instill intranasally
Arm/Group | Arm A (Rose Geranium in Sesame Oil Nasal Spray) | Arm B (Isotonic Nasal Saline) | Arm A Crossover | Arm B Crossover
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/53 | 0/2 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53 | 0/2 | 0/37
Other Adverse Events (participants affected / at risk) | 10/53 | 9/53 | 0/2 | 4/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Rose Geranium in Sesame Oil Nasal Spray) (N=53) | Arm B (Isotonic Nasal Saline) (N=53) | Arm A Crossover (N=2) | Arm B Crossover (N=37)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
White blood cell decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT04620369/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT04620369/ICF_001.pdf